CLINICAL TRIAL: NCT04055051
Title: An Observational Cohort Study of Long-Term Outcomes of Orthotopic Liver Transplantation in People With Hemophilia
Brief Title: ATHN 11: Liver Transplantation Outcomes Study
Acronym: HOT
Status: Completed | Type: Observational
Sponsor: American Thrombosis and Hemostasis Network (Network)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: ATHN 11: Liver Transplantation
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hemophilia A and B; Liver Transplantation
Keywords: Hemophilia A; Hemophilia B; Liver Transplantation; Quality of Life; Hemophilia Treatment Centers (HTCs)
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemophilia A and B Cases: No intervention. Only patients that have undergone a liver transplant per study eligibility are in this cohort.
- Hemophilia A and B Controls: No intervention. Comparable patients to those in Case cohort will be put in this cohort.

SUMMARY:
This study is designed as a multi-center, observational cohort study of participants with hemophilia A and B who have and have not undergone liver transplantation. Participants will be asked to complete health related quality of life questionnaires and provide medical history.

DETAILED DESCRIPTION:
At a time when gene therapy is becoming a reality for individuals with hemophilia A and B, little is known about long-term cures. Yet, there are few data to provide real life testing of the impact of long-term cures. Specifically, little is known about the relationship between factor level achieved with gene therapy and clinical outcomes or quality of life. The analogy to liver transplant is clear. There has been no systematic method to collect and analyze the long-term outcomes of liver transplantation in individuals with hemophilia. Previous efforts to access data through the United Network for Organ Sharing national database have been complicated by lack of identification of those with hemophilia. As most of the individuals with hemophilia who undergo liver transplantation receive care at a hemophilia treatment center (HTC), ATHN proposes to leverage its existing relationship with the HTCs to support HTC execution of this study.

ATHN, in collaboration with US Hemophilia Treatment Centers (HTCs), can provide the infrastructure and organization to support a longitudinal cohort study of subjects with congenital hemophilia who have and have not undergone liver transplantation. This cohort study will compare quality of life outcomes between cases that have undergone liver transplantation and controls that have not undergone liver transplantation. The study will determine if factor levels attained post-transplantation correlate with or predict improvement in quality of life measures.

The existence of ATHN and the ATHN System for clinical care and research provides an opportunity to observe a cohort of subjects after liver transplantation with facility. During the study period, it is predicted that sustained normalization in factor VIII or IX levels following liver transplantation improves clinical functioning and quality of life in adults with hemophilia A and B.

All study related contact will be timed to coincide with routine, scheduled care whenever possible. The study schedule will include:

Study enrollment - Study activities will begin after participant consent. Activities include the documentation of relevant medical history and the administration of quality of life (QoL) questionnaires.

Participants will be asked to complete health related (QoL) questionnaires and provide medical history. These questionnaires include:

1. Hemophilia Quality of Life Questionnaire for Adults (Haem-A-QoL): A quality of life questionnaire designed to asses health-related quality of life in adult patients with hemophilia. Domains include physical health, feelings, view of self, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, and partnership and sexuality.
2. Patient Reported Outcomes Measurement Information System (PROMIS-29): A quality of life questionnaire designed to assess physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity.
3. Hemophilia Orthotopic Liver Transplantation QoL Questionnaire (HOT): A quality of life questionnaire, adapted from a cancer survivorship tool, designed to assess adults with hemophilia who have received a liver transplant. Domains include physical well-being, psychological well-being, stress, anxiety, fear, work, family, relationships, and spiritual well-being.

ELIGIBILITY:
Inclusion Criteria

Participants who meet the following inclusion criteria are eligible for enrollment into the study:

1. Congenital hemophilia A or B of any severity, who have and have not undergone a liver transplant;
2. Age > 18; and
3. Sex assigned at birth was male

Exclusion Criteria

Participants who fall into any of the following exclusion criteria at the time of screening are not eligible for enrollment into the study:

1. Age <18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll a cohort of approximately 112 participants born with hemophilia who meet the eligibility criteria and are receiving care from one of approximately 12 participating HTCs. The participants will be approached for enrollment and matched 1:3 with age-, race-, ethnicity-matched controls (N=84) with hemophilia who have not undergone transplantation, for a total of 112 individuals with hemophilia who will compete quality of life questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (Haem-A-QoL) | 1 year
  Health related quality of life questionnaire Hemophilia Quality of Life Questionnaire for Adults (Haem-A-QoL): Domains include physical health, feelings, view of self, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, and partnership and sexuality.
  For comparing questionnaire scores between two cohorts, we could use a combined score of PROMIS-29, Haem-A-QoL, and HOT questionnaires rescaled in 0-100 or use each separate survey.
Quality of life (PROMIS-29) | 1 year
  Health related Quality of Life measured by the Patient Reported Outcome Measurement Information System (PROMIS-29) Profile measure physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity.
Quality of Life (HOT) | 1 year
  Hemophilia Orthotopic Liver Transplantation QoL Questionnaire (HOT) Domains include physical well-being, psychological well-being, stress, anxiety, fear, work, family, relationships and spiritual well-being.

SECONDARY OUTCOMES:
Clotting factor protein | 1year
  impact of sustained increase in clotting factor proteins (FVIII and FIX) levels after liver transplantation. The medical record will be accessed to record baseline hemophilia history including primary factor diagnosis and baseline factor level used to access disease severity, post-transplant factor levels and genotype.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Ragni, MD, MPH, Principal Investigator — University of Pittsburgh Medical Center
Locations (15):
- United States (15):
  - Orthopaedic Institute for Children Hemophilia Program, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center (IHTC), Indianapolis, Indiana
  - Maine Hemophilia and Thrombosis Center, Scarborough, Maine
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Comprehensive Hemophilia Center, Rochester, Minnesota
  - Mary M. Gooley Hemophilia Center, Inc., Rochester, New York
  - Comprehensive Hemophilia Treatment Center, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Medical Center Hemophilia Treatment Center, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Gulf States Hemophilia and Thrombophilia Center, Houston, Texas
  - Utah Center for Bleeding and Clotting Disorders, Salt Lake City, Utah
  - Hemophilia Outreach Center Green Bay, Green Bay, Wisconsin
  - Comprehensive Center for Bleeding Disorders, Milwaukee, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madeira CL, Layman ME, de Vera RE, Fontes PA, Ragni MV. Extrahepatic factor VIII production in transplant recipient of hemophilia donor liver. Blood. 2009 May 21;113(21):5364-5. doi: 10.1182/blood-2009-02-206979. No abstract available. PMID 19470440
- [Background] Subramanian A, Sulkowski M, Barin B, Stablein D, Curry M, Nissen N, Dove L, Roland M, Florman S, Blumberg E, Stosor V, Jayaweera DT, Huprikar S, Fung J, Pruett T, Stock P, Ragni M. MELD score is an important predictor of pretransplantation mortality in HIV-infected liver transplant candidates. Gastroenterology. 2010 Jan;138(1):159-64. doi: 10.1053/j.gastro.2009.09.053. Epub 2009 Sep 30. PMID 19800334
- [Background] Ragni MV, Moore CG, Soadwa K, Nalesnik MA, Zajko AB, Cortese-Hassett A, Whiteside TL, Hart S, Zeevi A, Li J, Shaikh OS; HHH Study Group. Impact of HIV on liver fibrosis in men with hepatitis C infection and haemophilia. Haemophilia. 2011 Jan;17(1):103-11. doi: 10.1111/j.1365-2516.2010.02366.x. Epub 2010 Aug 16. PMID 20722744
- [Background] Ragni MV, Devera ME, Roland ME, Wong M, Stosor V, Sherman KE, Hardy D, Blumberg E, Fung J, Barin B, Stablein D, Stock PG. Liver transplant outcomes in HIV+ haemophilic men. Haemophilia. 2013 Jan;19(1):134-40. doi: 10.1111/j.1365-2516.2012.02905.x. Epub 2012 Jul 5. PMID 22762561
- [Background] Terrault NA, Roland ME, Schiano T, Dove L, Wong MT, Poordad F, Ragni MV, Barin B, Simon D, Olthoff KM, Johnson L, Stosor V, Jayaweera D, Fung J, Sherman KE, Subramanian A, Millis JM, Slakey D, Berg CL, Carlson L, Ferrell L, Stablein DM, Odim J, Fox L, Stock PG; Solid Organ Transplantation in HIV: Multi-Site Study Investigators. Outcomes of liver transplant recipients with hepatitis C and human immunodeficiency virus coinfection. Liver Transpl. 2012 Jun;18(6):716-26. doi: 10.1002/lt.23411. PMID 22328294
- [Background] Aguero F, Rimola A, Stock P, Grossi P, Rockstroh JK, Agarwal K, Garzoni C, Barcan LA, Maltez F, Manzardo C, Mari M, Ragni MV, Anadol E, Di Benedetto F, Nishida S, Gastaca M, Miro JM; FIPSE/NIH HIVTR/NEAT023 Investigators. Liver Retransplantation in Patients With HIV-1 Infection: An International Multicenter Cohort Study. Am J Transplant. 2016 Feb;16(2):679-87. doi: 10.1111/ajt.13461. Epub 2015 Sep 28. PMID 26415077
- [Background] Mehta KD, Ragni MV. Bleeding and liver transplantation outcomes in haemophilia. Haemophilia. 2017 Mar;23(2):230-237. doi: 10.1111/hae.13104. Epub 2016 Nov 4. PMID 27813318
- [Background] Ragni MV, Humar A, Stock PG, Blumberg EA, Eghtesad B, Fung JJ, Stosor V, Nissen N, Wong MT, Sherman KE, Stablein DM, Barin B. Hemophilia Liver Transplantation Observational Study. Liver Transpl. 2017 Jun;23(6):762-768. doi: 10.1002/lt.24688. PMID 27935212
- [Background] Ragni MV, Nalesnik MA, Schillo R, Dang Q. Highly active antiretroviral therapy improves ESLD-free survival in HIV-HCV co-infection. Haemophilia. 2009 Mar;15(2):552-8. doi: 10.1111/j.1365-2516.2008.01935.x. PMID 19347994